CLINICAL TRIAL: NCT00327093
Title: Elaboration of a Model for Predicting Efficacy of Monoclonal Antibodies (Cetuximab and Bevacizumab) in Patients With Colorectal Cancer and Liver Metastases
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The scientific commitee decided to stop the inclusions and exploit the results.
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Jean-Alain CHAYVIALLE, Pr, Hospices Civils de Lyon
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-401
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2009-02

CONDITIONS: Colorectal Cancer; Neoplasm Metastasis
Keywords: Colorectal cancer,; immunohistochemistry,; monoclonal antibodies,; predictive model,; antiangiogenic agents,; medical imaging; Colorectal cancer with liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Cetuximab; Bevacizumab

ARMS (2):
- 1 (Experimental): Bevacizumab
  Interventions: Drug: bevacizumab
- 2 (Experimental): Cetuximab
  Interventions: Drug: cetuximab

INTERVENTIONS:
Drug: cetuximab — indication : second intention treatment
  Other Names: Erbitux
  Arms: 2
Drug: bevacizumab — Indication: first intention treatment
  Other Names: Avastin
  Arms: 1

SUMMARY:
Primary Objective: This trial is elaborating a model for rapidly predicting (day 21) the response to monoclonal antibodies anti-EGFR and anti-VEGF (cetuximab and bevacizumab) based on biological markers and/or functional imaging. The response to treatment is evaluated by the conventional method after 2 months (Response Evaluation Criteria in Solid Tumors [RECIST] criteria).

Secondary Objectives:

1. This trial is also analyzing the correlation between the magnitude of response to treatment at 2 months (stabilization or objective response, RECIST criteria) and that of response observed after 6 months of treatment.
2. The organisational objective is to develop a tumour bank of metastatic colorectal cancer.

Population: The population includes 252 male and female patients with metastatic colorectal cancer justifying the use of cetuximab or bevacizumab, with no heart disease.

Techniques: Computed tomography (CT scan), functional imaging (ultrasound with SonoVue); molecular imaging (positron emission tomography [PET] with fluorodeoxyglucose F18 [18-FDG]); and biology and pathology on microbiopsy of liver metastasis are used.

Outcome Criteria: The primary outcome is response to treatment with monoclonal antibodies according to RECIST criteria at two months.

Studied Factors:

Radiology:

1. CT scan: RECIST criteria (gold standard);
2. Ultrasound with SonoVue injection: 1 representative target (delay of contrast appearance, peak of rising, curve of increase and decrease of the signal, area under the curve, time of average transit).

Nuclear Medicine: PET scan and 18-FDG (standard uptake values [SUV])

Molecular Characterization of Tumors: p53 status; microsatellite instability (MSI) status; expression of oncogenes; EGFR status; VEGF status; determination of FcgammaRIIIA polymorphisms

Statistics:

1. Descriptive analyses;
2. Analysis of the appropriate threshold to measure: response to treatment by an ultrasound with SonoVue and by PET scan; correlation between response predicted by the ultrasound with SonoVue and the PET; conventional morphological CT at 2 months
3. Analysis of prognostic factors:

   1. Evaluation of the role of each prognostic factor (pathology and imaging) on response to treatment;
   2. Multivariate analysis of prognostic factors;
   3. Analysis of the prognostic power of early response at 2 months on the response observed after 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 18 years old
* Patients with colon or rectal carcinoma histologically proven
* Patients with metastases (synchronous or metachronous)
* Patients with associated extra-hepatic disease (asymptomatic primary tumor or extra-hepatic metastases)
* Performance status (World Health Organization [WHO]) = 0, 1, or 2
* Life expectancy >= 3 months
* Patients with normal haematological, kidney, and liver parameters (PNN > 1.5 x 10^9/L, platelets > 100 10^9/L, total bilirubin <= 1.25 x upper limit of normal (ULN), ASAT/ALAT <= 5 x ULN, creatinaemia <= 135 µmol/L (1.5 mg/dL)
* No cardiac or coronary insufficiency untreated
* At least 4 weeks between surgery and study beginning
* Patients can have a biopsy of the hepatic lesion identified by ultrasound.
* Informed consent signed.

Exclusion Criteria:

* Patients with symptomatic tumors (colon or rectal)
* Patients with others tumors not cured
* Patients who cannot be treated by 5-fluorouracil (5-FU) and/or irinotecan because of special medical conditions or other serious disease.
* Patients who participated in another clinical trial since less than 30 days
* Pregnancy or breast-feeding women
* Patients who cannot be treated because of active infection or other serious disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Elaboration of a predictive model, based on biological and functional imaging parameters, for the response to monoclonal antibodies as assessed through RECIST criteria 2 months after the beginning of treatment | at 7 weeks

SECONDARY OUTCOMES:
Correlation between the response at 2 months and that at 6 months of treatment (taking into account the therapeutic adjustments during the 6-month follow-up) | at 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Alain Chayvialle, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Jean-Alain Chayvialle, Lyon, France